CLINICAL TRIAL: NCT05616728
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Effects of EDP-235 in Non-hospitalized Adults With Mild or Moderate COVID-19
Brief Title: A Study to Evaluate EDP-235 in Non-hospitalized Adults With COVID-19
Acronym: SPRINT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EDP 235-101
Record Dates: First submitted 2022-11-09; First posted 2022-11-15 (Actual); Results first posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-05

CONDITIONS: COVID-19
Keywords: SARS-CoV-2, Standard Risk
MeSH Terms: conditions — COVID-19 | interventions — EDP-235

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- EDP-235 200mg (Experimental): Once a day orally for 5 days
  Interventions: Drug: EDP-235
- EDP-235 400mg (Experimental): Once a day orally for 5 days
  Interventions: Drug: EDP-235
- Placebo (Placebo Comparator): Once a day orally for 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EDP-235 — capsule
  Arms: EDP-235 200mg; EDP-235 400mg
Drug: Placebo — capsule
  Arms: Placebo

SUMMARY:
Study of EDP-235 in Non-hospitalized Adults with Mild or Moderate COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2 infection confirmed by positive test ≤24 hours before randomization
* COVID-19 symptom onset within 5 days prior to randomization and at least 2 signs/symptoms attributable to COVID-19 present and one of at least moderate severity at Screening

Exclusion Criteria:

* Prior SARS-CoV-2 infection <90 days before enrollment and/or received any COVID-19 vaccine dose <90 days before enrollment
* Has one or more conditions associated with high risk for severe COVID-19
* History of hospitalization for the medical treatment of COVID-19
* Currently hospitalized or anticipated need for hospitalization in the clinical opinion of the investigator
* Known medical history of active liver disease
* Receiving dialysis or have known moderate to severe renal impairment
* Suspected or confirmed concurrent active systemic infection other than COVID-19 that may interfere with the evaluation of response to the study drug
* Any comorbidity requiring hospitalization and/or surgery within 7 days before study entry, or that is considered life threatening within 30 days before study entry
* Known HIV infection with a HIV viral load greater than 400 copies/mL or medication for HIV treatment that is prohibited in this study based on medical history within 6 months before the screening visit
* History of hypersensitivity or other contraindication to any of the components of the study drug
* Has received or is expected to receive pre-exposure prophylactic SARS-CoV-2 mAb
* Has received or is expected to receive convalescent COVID-19 plasma
* Oxygen saturation of ≤93% on room air obtained at rest within 24 hours before randomization
* Participating in another interventional clinical study with an investigational agent or device, including those for COVID-19, within 30 days or five half-lives of the agent, whichever is longer, before signing the ICF
* Females who are pregnant or breastfeeding

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 231 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Inc, Study Director — Enanta Pharmaceuticals, Inc
Locations (23):
- United States (22):
  - Torrance Clinical Research Institute, Lomita, California
  - LA Universal Research Center, Inc., Los Angeles, California
  - MedBio Trials - Miami, Aventura, Florida
  - Doral Medical Research, Doral, Florida
  - Encore Medical Research - Hollywood, Hollywood, Florida
  - Universal Medical and Research Center, LLC, Hollywood, Florida
  - Advanced Research for Health Improvement, LLC, Immokalee, Florida
  - LCC Medical Research - Miami - ClinEdge - PPDS, Miami, Florida
  - USPA Advance Concept Medical Research Group. LLC, Miami, Florida
  - Continental Clinical Research, LLC, Miami, Florida
  - Dynamic Medical Research, LLC - Miami, Miami, Florida
  - BioClinical Research Alliance, Miami, Florida
  - D&H National Research Centers, Miami, Florida
  - Florida International Medical Research, Miami, Florida
  - C'A Medical Center Inc Research, Miami, Florida
  - Reed Medical Research, Miami, Florida
  - CDC Research Institute, LLC, Port Saint Lucie, Florida
  - Carolina Research Center, Shelby, North Carolina
  - Toledo Institute of Clinical Research, Toledo, Ohio
  - Trio Clinical Trials LLC, Houston, Texas
  - SMS Clinical Research, LLC, Mesquite, Texas
  - Epic Medical Research, Red Oak, Texas
- County Emergency Hospital, Cluj-Napoca, Cluj, Romania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EDP-235 200mg | EDP-235 400mg | Placebo
Started | 77 | 78 | 76
Completed | 75 | 74 | 74
Not Completed | 2 | 4 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Physician Decision | 1 | 1 | 1
Not completed — Other | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EDP-235 200mg | EDP-235 400mg | Placebo | Total
Number analyzed (Participants) | 77 | 78 | 76 | 231
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (13.02) | 44.8 (11.77) | 42.8 (11.80) | 43.7 (12.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 47 | 42 | 139
  Male | 27 | 31 | 34 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 74 | 73 | 71 | 218
  Not Hispanic or Latino | 3 | 5 | 5 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 5 | 9
  White | 73 | 75 | 70 | 218
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events as a Measure of Safety and Tolerability
Time Frame: Day 1 through Day 33
Measure: Number; unit: Number of Adverse Events
Arm/Group | EDP-235 200mg | EDP-235 400mg | Placebo
Number analyzed (Participants) | 77 | 78 | 76
Number of Adverse Events | 1 | 6 | 3

2. Secondary Outcome: Change From Baseline in SARS-CoV-2 RNA Viral Load
Time Frame: Day 3, Day 5, Day 9 and Day 14
Population: Only subjects with a value at both baseline and the specific post-baseline visit are included.
Measure: Mean (Standard Deviation); unit: Viral load (log10 TCID50/mL)
Arm/Group | EDP-235 200mg | EDP-235 400mg | Placebo
Number analyzed (Participants) | 62 | 67 | 61
Viral load (log10 TCID50/mL)
  Day 3 | -1.664 (1.9974) | -1.626 (2.0049) | -1.500 (1.8459)
  Day 5 | -3.048 (2.0395) | -3.465 (1.7871) | -3.340 (1.7956)
  Day 9 | -4.198 (1.8878) | -4.237 (1.6148) | -4.441 (1.5036)
  Day 14 | -4.611 (1.5681) | -4.715 (1.5728) | -4.757 (1.4700)

3. Secondary Outcome: Change From Baseline in Infectious SARS- CoV-2 Viral Load
Time Frame: Day 3, Day 5, Day 9 and Day 14
Population: Only subjects with a value at both baseline and the specific post-baseline visit are included.
Measure: Mean (Standard Deviation); unit: Viral load (log10 TCID50/mL)
Arm/Group | EDP-235 200mg | EDP-235 400mg | Placebo
Number analyzed (Participants) | 62 | 67 | 61
Viral load (log10 TCID50/mL)
  Day 3 | -0.743 (1.5220) | -0.836 (1.3531) | -0.705 (1.3627)
  Day 5 | -0.872 (1.4164) | -1.065 (1.1804) | -0.982 (1.3341)
  Day 9 | -0.926 (1.4611) | -1.111 (1.2072) | -1.018 (1.3479)
  Day 14 | -0.959 (1.4153) | -1.111 (1.2072) | -1.009 (1.3589)

4. Secondary Outcome: Proportion of Participants With COVID-19 Signs/Symptom Improvement
Time Frame: Day 1 through Day 33
Measure: Count of Participants; unit: Participants
Arm/Group | EDP-235 200mg | EDP-235 400mg | Placebo
Number analyzed (Participants) | 62 | 67 | 61
Participants | 56 | 61 | 51

5. Secondary Outcome: Change From Baseline in COVID-19 Signs/Symptom
Description: The total score is computed as the sum across all 14 COVID-19 symptom severity scores for each visit. Total scores range from 0 to 42; higher scores indicate more severe symptoms. For symptom score, 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe for each symptom.
Time Frame: Day 1 through Day 33
Population: Only subjects with a value at both baseline and the specific post-baseline visit are included.
Measure: Mean (Standard Deviation); unit: Total score
Arm/Group | EDP-235 200mg | EDP-235 400mg | Placebo
Number analyzed (Participants) | 62 | 67 | 61
Total score | -12.8 (5.94) | -14.0 (6.20) | -12.8 (4.93)

6. Secondary Outcome: Proportion of Participants With Medically Attended Visits for COVID-19
Time Frame: Day 1 through Day 33
Measure: Count of Participants; unit: Participants
Arm/Group | EDP-235 200mg | EDP-235 400mg | Placebo
Number analyzed (Participants) | 62 | 67 | 61
Participants | 0 | 0 | 0

7. Secondary Outcome: Proportion of Participants Requiring Hospitalization for COVID-19
Time Frame: Day 1 through Day 33
Measure: Count of Participants; unit: Participants
Arm/Group | EDP-235 200mg | EDP-235 400mg | Placebo
Number analyzed (Participants) | 62 | 67 | 61
Participants | 0 | 0 | 0

8. Secondary Outcome: Proportion of Participants All-cause Mortality
Time Frame: Day 1 through Day 33
Measure: Count of Participants; unit: Participants
Arm/Group | EDP-235 200mg | EDP-235 400mg | Placebo
Number analyzed (Participants) | 77 | 78 | 76
Participants | 0 | 0 | 0

9. Secondary Outcome: Proportion of Participants Who Require Hospitalization and Mechanical Ventilation
Time Frame: Day 1 through Day 33
Measure: Count of Participants; unit: Participants
Arm/Group | EDP-235 200mg | EDP-235 400mg | Placebo
Number analyzed (Participants) | 62 | 67 | 61
Participants | 0 | 0 | 0

10. Secondary Outcome: Mean Plasma PK Concentrations of EDP-235
Time Frame: Day 1 through Day 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | EDP-235 200mg | EDP-235 400mg
Number analyzed (Participants) | 70 | 76
ng/mL
  Study Day 1 Postdose | 571 (159) | 902 (108)
  Study Day 3 Predose | 1050 (95.8) | 2250 (70.0)
  Study Day 5 Predose | 1290 (79.4) | 2230 (69.0)

ADVERSE EVENTS:
Time Frame: Through day 33
Arm/Group | EDP-235 200mg | EDP-235 400mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/78 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/78 | 0/76
Other Adverse Events (participants affected / at risk) | 1/77 | 5/78 | 2/76
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EDP-235 200mg (N=77) | EDP-235 400mg (N=78) | Placebo (N=76)
Hepatotoxicity (Hepatobiliary disorders) | 1 | 1 | 0 — These were mild increases in transaminases that were asymptomatic and were not accompanied by increases in alkaline phosphatase or bilirubin.
Periorbital oedema (Eye disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Face oedema (General disorders) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-02-13): https://cdn.clinicaltrials.gov/large-docs/28/NCT05616728/Prot_002.pdf
  • Statistical Analysis Plan (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/28/NCT05616728/SAP_003.pdf